CLINICAL TRIAL: NCT02122796
Title: A Pilot Randomized Controlled Trial to Assess the Impact of Acupuncture on Post-mastectomy Pain, Nausea, Anxiety and Ability to Cope.
Brief Title: A Pilot Trial to Assess the Impact of Acupuncture on Post-mastectomy Pain, Nausea, Anxiety and Ability to Cope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S121301
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mastectomy; Acupuncture
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Two sessions of acupuncture, at least twelve hours apart, post-mastectomy.
  Interventions: Other: Acupuncture
- Standard of Care (No Intervention): Standard of care post-mastectomy.

INTERVENTIONS:
Other: Acupuncture — Acupuncture involves inserting thin, sterile needles into the skin at certain points in the body.
  Arms: Acupuncture

SUMMARY:
The purpose of the study is to compare the effect of acupuncture to the standard of care (control group) on pain, nausea, anxiety, ability to cope, costs and length of hospital stay in post-mastectomy patients at Abbott Northwestern Hospital.

DETAILED DESCRIPTION:
About 40 subjects will be participating in this study. Following qualification for the study, participants will be randomly assigned by chance to receive either acupuncture or to receive the standard of care without an integrative medicine session.

* One group will receive acupuncture after surgery. Acupuncture involves inserting thin, sterile needles at certain points on your body.
* The other group will receive the standard of care without an acupuncture session.

Before surgery participants will complete a demographics questionnaire. After surgery, participants will be visited in their hospital room by either an acupuncturist or another member of the research team. For those assigned to the acupuncture group, participants will receive up to two sessions of acupuncture, at least twelve hours apart. For those assigned to the control group, a research team member will visit the participant in their room up to two times, at least twelve hours apart. During those visits, participants will be asked about pain, nausea, anxiety, and ability to cope at the beginning and end of each treatment or visit.

Additional information will be gathered from participants hospital charts, such as the type of surgery that was performed, length of hospital stay, and the costs associated with the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years or older
* Undergoing mastectomy surgery

Exclusion Criteria:

* Non-English speaking
* Pregnant
* Also undergoing an oophorectomy, TRAM or Latissimus flap surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Visit 1
Arm/Group | Acupuncture | Standard of Care
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Acupuncture | Standard of Care
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Standard of Care | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.74 (9.41) | 62.47 (11.47) | 57.52 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Number; unit: participants]
  <9th Grade | 0 | 0 | 0
  9th to 12th Grade | 0 | 1 | 1
  High School Graduate | 4 | 3 | 7
  Some College or Associate Degree | 5 | 7 | 12
  Bachelor's Degree or Higher | 6 | 4 | 10
Employment Status [Number; unit: participants]
  Full-time | 8 | 4 | 12
  Part-time | 3 | 3 | 6
  Homemaker | 2 | 2 | 4
  Retired | 2 | 6 | 8
  Other | 0 | 0 | 0
Family Income [Number; unit: participants]
  <$24,999 | 0 | 2 | 2
  $25,000-39,999 | 1 | 0 | 1
  $40,000-54,999 | 4 | 1 | 5
  $55,000-74,999 | 2 | 3 | 5
  $75,000 or more | 8 | 7 | 15
  Unknown | 0 | 2 | 2
Marital Status [Number; unit: participants]
  Married | 12 | 12 | 24
  Living in marriage-like relationship | 0 | 0 | 0
  Divorced/separated | 2 | 3 | 5
  Widowed | 1 | 0 | 1
  Never married | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Eligible Compared to the Number Approached and Enrolled
Description: Feasibility will be measured by the number of patients eligible for enrollment, the number approached, the number consented, and the final sample with completed data. The study population will be described in terms of demographics and background characteristics collected on the enrollment questionnaire.
Time Frame: One year
Population: A total of 252 women were scheduled to receive a unilateral or bilateral mastectomy during the study period. Of those, 61 were eligible for study participation, and there were 30 women who provided consent and were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Undergoing Mastectomy Surgery: Number of individuals having mastectomy surgery who were approached for participation in the trial
Arm/Group | Patients Undergoing Mastectomy Surgery
Number analyzed (Participants) | 252
Participants
  Elligible | 61
  Approached | 252
  Consented | 30
  Declined | 31
  Final Sample with complete data | 26

2. Secondary Outcome: Change in Pain Post Intervention
Description: Change in pain on a single question 11-point Numeric Rating Scale (NRS) where 0 equals no pain and 10 equals most severe pain. The score is derived by subtracting the pre-intervention score from the post-intervention score within the same day (e.g. Post-Pain Day 1 - Pre-Pain Day 1). A lower score indicates better outcomes. Outcomes were obtained on both post-op Day 1 and Day 2.
Time Frame: Participants will be followed on post operations day 1 and 2 of their hospital stay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 12 | 14
units on a scale
  Visit 1 Mean Change in Pain | -1.47 (1.06) | -0.07 (1.67)
  Visit 2 Mean Change in Pain | -1.50 (0.97) | -0.43 (1.02)
Statistical Analysis 1: Comparison: Acupuncture vs Standard of Care; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — Means of pre- and post-treatment measurements were compared using paired, two-sided Student's t tests. P values were calculated comparing acupuncture and control mean change scores using unpaired two-sided Student's t tests; P values were calculated comparing acupuncture and control mean change scores using unpaired two-sided Student's t tests

3. Secondary Outcome: Change in Anxiety Post Intervention
Description: Change in anxiety on a single question 11-point Numeric Rating Scale (NRS) where 0 equals no anxiety and 10 equals most severe anxiety. The score is derived by subtracting the pre-intervention score from the post-intervention score within the same day (e.g. Post-Anxiety Day 1 - Pre-Anxiety Day 1). A lower score indicates better outcomes. Outcomes were obtained on both post-op Day 1 and Day 2.
Time Frame: Participants will be followed on post operations day 1 and 2 of their hospital stay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 12 | 14
units on a scale
  Visit 1 Change in Anxiety | -1.33 (1.59) | 0.53 (2.88)
  Visit 2 Change in Anxiety | -0.90 (1.45) | 0.14 (1.03)
Statistical Analysis 1: Comparison: Acupuncture vs Standard of Care; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Nausea Post Intervention
Description: Change in nausea on a single question 11-point Numeric Rating Scale (NRS) where 0 equals no nausea and 10 equals most severe nausea. The score is derived by subtracting the pre-intervention score from the post-intervention score within the same day (e.g. Post-Nausea Day 1 - Pre-Nausea Day 1). A lower score indicates better outcomes. Outcomes were obtained on both post-op Day 1 and Day 2.
Time Frame: Participants will be followed on post operations day 1 and 2 of their hospital stay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 12 | 14
units on a scale
  Visit 1 Change in Nausea | -1.53 (2.70) | 0.73 (1.75)
  Visit 2 Change in Nausea | -0.50 (1.27) | -0.29 (1.38)

5. Secondary Outcome: Change in Ability to Cope Post Intervention
Description: Change in ability to cope on a single question 11-point Numeric Rating Scale (NRS) where 0 equals absence of an ability to cope and 10 equals complete ability to cope. The score is derived by subtracting the pre-intervention score from the post-intervention score within the same day (e.g. Post-Coping Day 1 - Pre-Coping Day 1). . A higher score indicates better outcomes. Outcomes were obtained on both post-op Day 1 and Day 2.
Time Frame: Participants will be followed on post operations day 1 and 2 of their hospital stay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Standard of Care
Number analyzed (Participants) | 12 | 14
units on a scale
  Visit 1 Change in Ability to Cope | 1.87 (2.97) | -0.47 (1.36)
  Visit 2 Change in Ability to Cope | 0.30 (3.06) | 0.07 (0.47)
Statistical Analysis 1: Comparison: Acupuncture vs Standard of Care; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Arm/Group | Acupuncture | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes